CLINICAL TRIAL: NCT06830174
Title: Network Targeted Transcranial Direct Current Stimulation (tDCS) as a Treatment for Laryngeal Dystonia (LD)
Brief Title: tDCS for Laryngeal Dystonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Spasmodic Dysphonia Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000032414
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Laryngeal Dystonia
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Masking Description: Subjects and staff will be blind during the study and that subjects will be told of their assignment at the follow-up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Laryngeal Dystonia (LD) tDCS (Experimental): Adductor, Abductor and Mixed type LD with clinical evaluation of LD or with proof of LD diagnosis
  Interventions: Device: Starstim system

INTERVENTIONS:
Device: Starstim system — Transcranial direct current stimulation (tDCS)

SUMMARY:
This project will apply transcranial direct current stimulation (tDCS) to multiple brain areas to evaluate the effects as a potential treatment for laryngeal dystonia (formerly spasmodic dysphonia).

DETAILED DESCRIPTION:
Baseline neuroimaging data will be acquired from all participants via MRI, EEG. Each participant will be seen for multiple testing sessions over a five day period. LD participants will undergo the neuromodulation (HD-tDCS Stimulation) for twenty minutes while engaged in watching videos/movies or performing a word production task.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be clinically evaluated for the diagnosis of LD or have the proof of LD diagnosis. (Not applicable for control participants)
* No other known or history of speech, voice disorder other than LD.
* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Must not be pregnant.

Exclusion Criteria:

* All individuals who do not meet the above mentioned criteria are excluded from the study.
* Subjects with a history of epilepsy or depression or is claustrophobic.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cepstral peak prominence (CPP) | daily on Day 1-Day 5
  Cepstral peak prominence (CPP) as a robust objective measure of voice quality in the active, sham and no stimulation conditions.
Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) | daily on Day 1-Day 5
  Its primary purpose is to describe the severity of auditory-perceptual attributes of a voice problem, in a way that can be communicated among clinicians

CONTACTS AND LOCATIONS:
Overall Officials: Nabin Koirala, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Investigators do not have consent for patients for sharing their data yet, if that changes, de-identified data will be shared.